CLINICAL TRIAL: NCT05326191
Title: First-trimester Placental Ultrasound Study (First PLUS): an Observational Cohort Study to Assess the Clinical Utility of the OxNNet Toolkit for the Prediction of Adverse Pregnancy Outcomes.
Brief Title: First-trimester Placental Ultrasound Study
Acronym: First PLUS
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: University of Oxford (Other); Fetal Medicine Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 22/WM/0039
Record Dates: First submitted 2022-03-15; First posted 2022-04-13 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Fetal Growth Complications; Pregnancy Complications
Keywords: Ultrasound; Fetal Growth; Pregnancy
MeSH Terms: conditions — Pregnancy Complications | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — All study interventions/procedures will happen during the participants routine clinic visit in which they will receive their routine Ultrasound scan, followed by an additional research scan, which will take approximately 2-3 minutes. A blood sample will also be taken from participants as part of their routine pregnancy care. Residual blood from the same sample will be used to conduct an additional test to quantify Placental Growth Factor (PlGF). Participants will also be asked questions about their relevant medical history and demographic data which is also routinely collected as part of their pregnancy record.

SUMMARY:
An observational cohort study to assess the clinical utility of the OxNNet Toolkit for the prediction of adverse pregnancy outcomes.

DETAILED DESCRIPTION:
The First PLUS study is a single centre, prospective, observational study recruiting 4000 women from The Harris Birthright Centre, which provides ultrasound scanning for all women who would attend King's College Hospital NHS Foundation Trust for their pregnancy care.

This study aims to develop a tool to provide reliable measurements of placental size and estimate the blood flow within the placenta during the first trimester of pregnancy. These metrics hope to develop a screening tool for fetal growth restriction (FGR), which is a condition in which a baby fails to grow to its full potential and can cause adverse pregnancy outcomes and is the single most common cause of stillbirth. This devastating outcome could potentially be reduced by stratifying pregnancies into high risk, allowing women to undergo additional monitoring and limiting clinician resource to those in need of it most. Stillbirth is also a serious adverse pregnancy outcome that NHS England is looking to reduce the rate of as part of their long-term plan.

Women 18 years of age or older, attending their first trimester scan during 11-14 weeks of pregnancy, who has a viable pregnancy with no more than one baby with no major defects identified during the scan will be eligible to take part.

The study will take place over 24 months and participants will undergo a single study visit in which their demographics and routine medical history will be recorded, an additional research ultrasound scan will be conducted alongside their routine scan, and blood from a sample taken as part of routine care will be used to assess the level of Placental Growth Factor (PlGF). Participants will then be followed up until the completion of their pregnancy via their pregnancy records (remote follow up) and the outcome of their pregnancy will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* 18 years of age, or older
* Presenting for first-trimester combined test screening between 11+0 and 13+6 weeks of pregnancy
* Participant is willing and able to give informed consent for participation in the investigation.
* Able to understand written or verbal English and able to access methods of translation.
* In the opinion of the investigator, the participant is not at risk or under stress or limited in their ability to participate in the study activities.

Exclusion Criteria:

* Participant with a multiple pregnancy (more than one viable fetus) discovered at the scan
* Participant with a non-viable pregnancy discovered at the scan (no detectable heartbeat)
* Pregnancies with major defects identified during 11+0 to13+6 week scan
* Any pregnancy subsequently found to be chromosomally abnormal as a result of either prenatal or postnatal testing

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women attending the Fetal Medicine Foundation for their first-trimester screening scan
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Fetal Growth restriction (FGR) | 24 months
  Fetal Growth restriction (FGR) defined according to the ISUOG Delphi consensus guidelines for diagnosis of FGR, at the time of delivery.

SECONDARY OUTCOMES:
Small for Gestational Age (GSA) | 24 months
  Defined if <10 centile on population-based centiles or <10th centile on customised centiles, at the time of delivery.
Pre-eclampsia (with, and without, severe features) | 24 months
  Defined by the ACOG guidelines for hypertensive disorders of pregnancy:
  * Pre-term pre-eclampsia (delivery <37 weeks)
  * Late onset pre-eclampsia (delivery ≥37 weeks)
Gestational hypertension (PIH) | 24 months
  Defined by the ACOG guidelines for hypertensive disorders of pregnancy:
  * Pre-term gestational hypertension (delivery <37 weeks)
  * Late onset gestational hypertension (delivery ≥37 weeks)
Haemolysis, elevated liver enzymes and low platelets (HELLP) syndrome | 24 months
  Defined by the ACOG guidelines for hypertensive disorders of pregnancy:
  * Pre-term HELLP (delivery <37 weeks)
  * Late onset HELLP (delivery ≥37 weeks) Pre-term pre-eclampsia (delivery <37 weeks)
Eclampsia | 24 months
  Defined by the ACOG guidelines for hypertensive disorders of pregnancy(22)
  * Pre-term eclampsia (delivery <37 weeks)
  * Late onset eclampsia (delivery ≥37 weeks)
Gestational diabetes | 24 months
  Defined as fasting plasma glucose level ≥5.6 mmol/L and/or 2-h plasma glucose level ≥7.8 mmol/L after ingestion of 75g oral glucose.
Preterm Birth | 24 months
  Birth ≥24+0 weeks <37+0 weeks
Miscarriage | 24 months
  Live fetus at the first-trimester ultrasound scan but subsequent in utero fetal death or delivery <24+0 weeks
Stillbirth | 24 months
  Baby born with no signs of life at ≥24+0 weeks' gestation
Neonatal death | 24 months
  Baby born alive but dies within the first 28 days of life
Neonatal morbidity | 24 months
  * Neonatal intensive care unit admission and length of stay
  * Neonatal ventilation - defined as need of positive pressure (CPAP, NCPAP or intubation)
  * Respiratory distress syndrome - defined as need of ventilation with or without surfactant
  * Intraventricular haemorrhage (IVH) grade II or above - defined as bleeding into the ventricles
  * Neonatal sepsis confirmed bacteraemia in cultures
  * Anaemia - defined as low haemoglobin and / or haematocrit requiring blood transfusion
  * Necrotizing enterocolitis requiring surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kypros Nicolaides, BSc, MMBS, Principal Investigator — Fetal Medicine Foundation
Locations (1):
- King's College Hospital NHS, Fetal Medicine Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvesen K, Lees C, Abramowicz J, Brezinka C, Ter Haar G, Marsal K; Board of International Society of Ultrasound in Obstetrics and Gynecology (ISUOG). ISUOG statement on the safe use of Doppler in the 11 to 13 +6-week fetal ultrasound examination. Ultrasound Obstet Gynecol. 2011 Jun;37(6):628. doi: 10.1002/uog.9026. No abstract available. PMID 21618313
- [Background] Froen JF, Cacciatore J, McClure EM, Kuti O, Jokhio AH, Islam M, Shiffman J; Lancet's Stillbirths Series steering committee. Stillbirths: why they matter. Lancet. 2011 Apr 16;377(9774):1353-66. doi: 10.1016/S0140-6736(10)62232-5. PMID 21496915
- [Background] Campbell HE, Kurinczuk JJ, Heazell A, Leal J, Rivero-Arias O. Healthcare and wider societal implications of stillbirth: a population-based cost-of-illness study. BJOG. 2018 Jan;125(2):108-117. doi: 10.1111/1471-0528.14972. Epub 2017 Dec 14. PMID 29034559
- [Background] Cousens S, Blencowe H, Stanton C, Chou D, Ahmed S, Steinhardt L, Creanga AA, Tuncalp O, Balsara ZP, Gupta S, Say L, Lawn JE. National, regional, and worldwide estimates of stillbirth rates in 2009 with trends since 1995: a systematic analysis. Lancet. 2011 Apr 16;377(9774):1319-30. doi: 10.1016/S0140-6736(10)62310-0. PMID 21496917
- [Background] Pillay T, Modi N, Rivero-Arias O, Manktelow B, Seaton SE, Armstrong N, Draper ES, Dawson K, Paton A, Ismail AQT, Yang M, Boyle EM. Optimising neonatal service provision for preterm babies born between 27 and 31 weeks gestation in England (OPTI-PREM), using national data, qualitative research and economic analysis: a study protocol. BMJ Open. 2019 Aug 22;9(8):e029421. doi: 10.1136/bmjopen-2019-029421. PMID 31444186
- [Background] Monier I, Blondel B, Ego A, Kaminiski M, Goffinet F, Zeitlin J. Poor effectiveness of antenatal detection of fetal growth restriction and consequences for obstetric management and neonatal outcomes: a French national study. BJOG. 2015 Mar;122(4):518-27. doi: 10.1111/1471-0528.13148. Epub 2014 Oct 27. PMID 25346493
- [Background] Looney P, Stevenson GN, Nicolaides KH, Plasencia W, Molloholli M, Natsis S, Collins SL. Fully automated, real-time 3D ultrasound segmentation to estimate first trimester placental volume using deep learning. JCI Insight. 2018 Jun 7;3(11):e120178. doi: 10.1172/jci.insight.120178. eCollection 2018 Jun 7. PMID 29875312
- [Background] Looney P, Yin Y, Collins SL, Nicolaides KH, Plasencia W, Molloholli M, Natsis S, Stevenson GN. Fully Automated 3-D Ultrasound Segmentation of the Placenta, Amniotic Fluid, and Fetus for Early Pregnancy Assessment. IEEE Trans Ultrason Ferroelectr Freq Control. 2021 Jun;68(6):2038-2047. doi: 10.1109/TUFFC.2021.3052143. Epub 2021 May 25. PMID 33460372
- [Background] Yin Y, Looney P, Collins SL. Standardization of blood flow measurements by automated vascular analysis from power Doppler ultrasound scan. Proc SPIE Int Soc Opt Eng. 2020 Feb;11314:113144C. doi: 10.1117/12.2549349. Epub 2020 Mar 16. No abstract available. PMID 33132475
- [Background] Welsh AW, Fowlkes JB, Pinter SZ, Ives KA, Owens GE, Rubin JM, Kripfgans OD, Looney P, Collins SL, Stevenson GN. Three-dimensional US Fractional Moving Blood Volume: Validation of Renal Perfusion Quantification. Radiology. 2019 Nov;293(2):460-468. doi: 10.1148/radiol.2019190248. Epub 2019 Oct 1. PMID 31573404
- [Background] Barker DJ, Thornburg KL. Placental programming of chronic diseases, cancer and lifespan: a review. Placenta. 2013 Oct;34(10):841-5. doi: 10.1016/j.placenta.2013.07.063. Epub 2013 Aug 2. PMID 23916422
- [Background] Barker DJP. Fetal origins of cardiovascular disease. Ann Med. 1999;31(sup1):3-6. doi: 10.1080/07853890.1999.11904392. PMID 28850284
- [Background] Barker DJ. Adult consequences of fetal growth restriction. Clin Obstet Gynecol. 2006 Jun;49(2):270-83. doi: 10.1097/00003081-200606000-00009. PMID 16721106
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Mosimann B, Pfiffner C, Amylidi-Mohr S, Risch L, Surbek D, Raio L. First trimester combined screening for preeclampsia and small for gestational age - a single centre experience and validation of the FMF screening algorithm. Swiss Med Wkly. 2017 Aug 25;147:w14498. doi: 10.4414/smw.2017.14498. eCollection 2017. PMID 28871576
- [Background] Collins SL, Birks JS, Stevenson GN, Papageorghiou AT, Noble JA, Impey L. Measurement of spiral artery jets: general principles and differences observed in small-for-gestational-age pregnancies. Ultrasound Obstet Gynecol. 2012 Aug;40(2):171-8. doi: 10.1002/uog.10149. PMID 22102536
- [Background] Collins SL, Welsh AW, Impey L, Noble JA, Stevenson GN. 3D fractional moving blood volume (3D-FMBV) demonstrates decreased first trimester placental vascularity in pre-eclampsia but not the term, small for gestation age baby. PLoS One. 2017 Jun 1;12(6):e0178675. doi: 10.1371/journal.pone.0178675. eCollection 2017. PMID 28570600
- [Background] Wareing M, Myers JE, O'Hara M, Baker PN. Sildenafil citrate (Viagra) enhances vasodilatation in fetal growth restriction. J Clin Endocrinol Metab. 2005 May;90(5):2550-5. doi: 10.1210/jc.2004-1831. Epub 2005 Feb 15. PMID 15713717
- [Background] Cottrell E, Tropea T, Ormesher L, Greenwood S, Wareing M, Johnstone E, Myers J, Sibley C. Dietary interventions for fetal growth restriction - therapeutic potential of dietary nitrate supplementation in pregnancy. J Physiol. 2017 Aug 1;595(15):5095-5102. doi: 10.1113/JP273331. Epub 2017 Feb 27. PMID 28090634
- [Background] Dilworth MR, Andersson I, Renshall LJ, Cowley E, Baker P, Greenwood S, Sibley CP, Wareing M. Sildenafil citrate increases fetal weight in a mouse model of fetal growth restriction with a normal vascular phenotype. PLoS One. 2013 Oct 30;8(10):e77748. doi: 10.1371/journal.pone.0077748. eCollection 2013. PMID 24204949
- [Background] Jones TB, Price RR, Gibbs SJ. Volumetric determination of placental and uterine growth relationships from B-mode ultrasound by serial area-volume determinations. Invest Radiol. 1981 Mar-Apr;16(2):101-6. doi: 10.1097/00004424-198103000-00005. PMID 7216699
- [Background] Collins SL, Stevenson GN, Noble JA, Impey L. Rapid calculation of standardized placental volume at 11 to 13 weeks and the prediction of small for gestational age babies. Ultrasound Med Biol. 2013 Feb;39(2):253-60. doi: 10.1016/j.ultrasmedbio.2012.09.003. Epub 2012 Dec 4. PMID 23219036
- [Background] Law LW, Leung TY, Sahota DS, Chan LW, Fung TY, Lau TK. Which ultrasound or biochemical markers are independent predictors of small-for-gestational age? Ultrasound Obstet Gynecol. 2009 Sep;34(3):283-7. doi: 10.1002/uog.6455. PMID 19670336
- [Background] Hafner E, Metzenbauer M, Hofinger D, Stonek F, Schuchter K, Waldhor T, Philipp K. Comparison between three-dimensional placental volume at 12 weeks and uterine artery impedance/notching at 22 weeks in screening for pregnancy-induced hypertension, pre-eclampsia and fetal growth restriction in a low-risk population. Ultrasound Obstet Gynecol. 2006 Jun;27(6):652-7. doi: 10.1002/uog.2641. PMID 16514618
- [Background] Farina A. Systematic review on first trimester three-dimensional placental volumetry predicting small for gestational age infants. Prenat Diagn. 2016 Feb;36(2):135-41. doi: 10.1002/pd.4754. Epub 2016 Jan 19. PMID 26618611
- [Background] Stevenson GN, Collins SL, Ding J, Impey L, Noble JA. 3-D Ultrasound Segmentation of the Placenta Using the Random Walker Algorithm: Reliability and Agreement. Ultrasound Med Biol. 2015 Dec;41(12):3182-93. doi: 10.1016/j.ultrasmedbio.2015.07.021. Epub 2015 Sep 1. PMID 26341043
- [Background] Cheong KB, Leung KY, Li TK, Chan HY, Lee YP, Tang MH. Comparison of inter- and intraobserver agreement and reliability between three different types of placental volume measurement technique (XI VOCAL, VOCAL and multiplanar) and validity in the in-vitro setting. Ultrasound Obstet Gynecol. 2010 Aug;36(2):210-7. doi: 10.1002/uog.7609. PMID 20201116
- [Background] RONNEBERGER O, FISCHER P, BROX T. U-Net: Convolutional Networks for Biomedical Image Segmentation. International Conference on Medical Image Computing and Computer-Assisted Intervention 2015;Springer:234-41.
- [Background] Pijnenborg R, Vercruysse L, Hanssens M. The uterine spiral arteries in human pregnancy: facts and controversies. Placenta. 2006 Sep-Oct;27(9-10):939-58. doi: 10.1016/j.placenta.2005.12.006. Epub 2006 Feb 20. PMID 16490251
- [Background] Huang YH, Chen JH, Chang YC, Huang CS, Moon WK, Kuo WJ, Lai KJ, Chang RF. Diagnosis of solid breast tumors using vessel analysis in three-dimensional power Doppler ultrasound images. J Digit Imaging. 2013 Aug;26(4):731-9. doi: 10.1007/s10278-012-9556-5. PMID 23296913
- [Background] Huang SF, Chang RF, Moon WK, Lee YH, Chen DR, Suri JS. Analysis of tumor vascularity using three-dimensional power Doppler ultrasound images. IEEE Trans Med Imaging. 2008 Mar;27(3):320-30. doi: 10.1109/TMI.2007.904665. PMID 18334428
- [Background] Shia WC, Chen DR, Huang YL, Wu HK, Kuo SJ. Effectiveness of evaluating tumor vascularization using 3D power Doppler ultrasound with high-definition flow technology in the prediction of the response to neoadjuvant chemotherapy for T2 breast cancer: a preliminary report. Phys Med Biol. 2015 Oct 7;60(19):7763-78. doi: 10.1088/0031-9155/60/19/7763. PMID 26393306
- [Background] LEE TC, KASHYAP RL, CHU CN. Building Skeleton Models via 3-D Medial Surface Axis Thinning Algorithms. CVGIP: Graphical Models and Image Processing 1994;56:462-78
- [Background] VIDELA A, LIN C-L, MILLER JD. Watershed Functions Applied to a 3D Image Segmentation Problem for the Analysis of Packed Particle Beds. Particle & Particle Systems Characterization 2006; 23: 237-45
- [Background] Rubin JM, Adler RS, Fowlkes JB, Spratt S, Pallister JE, Chen JF, Carson PL. Fractional moving blood volume: estimation with power Doppler US. Radiology. 1995 Oct;197(1):183-90. doi: 10.1148/radiology.197.1.7568820.
- [Background] Yen PL, Wu HK, Tseng HS, Kuo SJ, Huang YL, Chen HT, Chen DR. Vascular morphologic information of three-dimensional power Doppler ultrasound is valuable in the classification of breast lesions. Clin Imaging. 2012 Jul-Aug;36(4):267-71. doi: 10.1016/j.clinimag.2011.11.012. Epub 2012 Jun 8. PMID 22726963
- [Background] CHIAO RY, BASHFORD GR, FEILEN MP, ANDREWS-OWEN C. Flash Artifact Suppression in Two-Dimensional Ultrasound Imaging. USA, 2004 (vol U. S. Patent No. 6,760,486.).
- [Background] Looney PT, Stevenson GN, Collins SL. 3D ultrasound file reading and coordinate transformations. J Open Source Softw. 2019;4(33):1063. doi: 10.21105/joss.01063. Epub 2019 Jan 11. PMID 31745534
- [Background] SUR F. An a-contrario approach to quasi-periodic noise removal2015 IEEE International Conference on Image Processing (ICIP), 2015
- [Background] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Background] Plasencia W, Akolekar R, Dagklis T, Veduta A, Nicolaides KH. Placental volume at 11-13 weeks' gestation in the prediction of birth weight percentile. Fetal Diagn Ther. 2011;30(1):23-8. doi: 10.1159/000324318. Epub 2011 Jun 23. PMID 21701132
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Riley RD, Snell KI, Ensor J, Burke DL, Harrell FE Jr, Moons KG, Collins GS. Minimum sample size for developing a multivariable prediction model: PART II - binary and time-to-event outcomes. Stat Med. 2019 Mar 30;38(7):1276-1296. doi: 10.1002/sim.7992. Epub 2018 Oct 24. PMID 30357870
- [Background] Zhan Y, Shen D, Zeng J, Sun L, Fichtinger G, Moul J, Davatzikos C. Targeted prostate biopsy using statistical image analysis. IEEE Trans Med Imaging. 2007 Jun;26(6):779-88. doi: 10.1109/TMI.2006.891497. PMID 17679329